CLINICAL TRIAL: NCT00162357
Title: Cardiolite-406; A Phase IV Open-Label, Randomized, Multi-Center Trial To Evaluate The Ability of Cardiolite Stress MPI to Detect Asymptomatic Restenosis in Diabetic Patients Who Have Undergone Percutaneous Coronary Intervention
Brief Title: Post-PCI:Cardiac Imaging in Patients With Diabetes to Detect Coronary Artery Blockages Previously Opened by Angioplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lantheus Medical Imaging (Industry)
Responsible Party: Qi Zhu, MD Sr. Medical Director, Lantheus Medical Imaging
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CARDIOLITE-406
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Diabetes Mellitus, Type 2; Coronary Restenosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Restenosis | interventions — Technetium Tc 99m Sestamibi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Technetium Tc99m Sestamibi

SUMMARY:
The purpose of this clinical research study is determine if patients with diabetes that have undergone previous opening of a heart blockage may have a blockage that is not causing any symptoms that may be detected by imaging with Cardiolite.

ELIGIBILITY:
Inclusion Criteria:

* Type II Diabetes on medication & angioplasty within the past 6 months.

Exclusion Criteria:

* Myocardial infarction or repeat angioplasty with the past 5 months.
* Unable to perform exercise or pharmacologic stress test.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2004-04; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Evaluate symptom-free heart blockages that develop following initial opening in patients with Type II diabetes mellitus based on Cardiolite imaging

SECONDARY OUTCOMES:
Determine how often symptom-free heart blockages occur 5-6 months after opening in patients with Type II diabetes mellitus
Examine the relative value of ejection fraction, summed stress, rest, and difference MPI scores for identifying patients with cardiac events during 18 month follow-up.
Compare patient hospital and out-patient cost for cardiac care for each group of patients (MPI versus standard care).

CONTACTS AND LOCATIONS:
Overall Officials: Qi Zhu, MD, Study Director — Lantheus Medical Imaging
Locations (8):
- United States (7):
  - Local Institution, Hartford, Connecticut
  - Local Institution, Waterbury, Connecticut
  - Local Institution, Grand Rapids, Michigan
  - Local Institution, Roslyn, New York
  - Local Institution, Burlington, Vermont
  - Local Institution, Roanoke, Virginia
  - Local Institution, Wausau, Wisconsin
- Local Institution, San Juan, Puerto Rico